CLINICAL TRIAL: NCT03924011
Title: The Use of Photobiomodulation Therapy for the Prevention of Acute Radiodermatitis in Breast Cancer Patients: a Multicentre, Randomized, Placebo-controlled Trial
Brief Title: Photobiomodulation Therapy for the Prevention of Acute Radiodermatitis in Breast Cancer Patients Undergoing Radiotherapy
Acronym: LABRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Prof. dr. Jeroen Mebis, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Labra-001
Record Dates: First submitted 2019-03-11; First posted 2019-04-23 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Radiodermatitis; Breast Cancer
Keywords: Radiodermatitis; Breast cancer; Radiotherapy; Photobiomodulation therapy; Low-level light therapy; Skin diseases; Radiation injuries; Wounds and injuries; Oncology
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms; Skin Diseases; Radiation Injuries; Wounds and Injuries; Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Receives sham laser (2x/week) in combination with standard skin care starting from day 1 of radiotherapy
  Interventions: Device: Sham laser
- Treatment group (Experimental): Receives PBMT (2x/week) in combination with standard skin care starting from day 1 of radiotherapy
  Interventions: Device: Photobiomodulation therapy (PBMT)

INTERVENTIONS:
Device: Photobiomodulation therapy (PBMT) — PBMT sessions will be planned 2x/week after RT.
  Other Names: Low-level light therapy (LLLT)
  Arms: Treatment group
Device: Sham laser — Sham laser sessions will be applied 2x/week after RT.
  Arms: Control group

SUMMARY:
Radiodermatitis (RD), an inflammatory skin reaction, occurs in more than 90 percent of cancer patients treated with radiotherapy (RT). This is the result of the radiation causing damage to the epidermal basal skin stem cells. Based on the severity of the skin symptoms, acute RD can be categorized into four grades ranging from red and dry skin to moist desquamation, necrosis, and eventually ulceration. Acute RD can be distressing, negatively influencing the patients' quality of life (QOL). In cases of severe RD, RT might be interrupted, affecting the treatment outcome.

Currently, there is no generally accepted treatment available for RD. As such, the standard skincare treatment is hospital dependent. Photobiomodulation therapy (PBMT) can offer a solution, since the therapeutic use of (infra)red light induces photochemical reactions in the target cells, stimulating repair and healing processes, and reducing pain and inflammation.

Previous studies using PBMT to prevent RD showed promising results. However, these beneficial results need to be validated in a larger breast cancer patient population receiving an alternative RT regimen. The study hypothesizes that PBMT is a safe and effective strategy to prevent worsening of acute RD grade two or higher in breast cancer patients undergoing RT. The primary objective is to measure the degree of acute RD to detect changes during and after RT. Second, the patients' QOL and pain will be assessed. Finally, the third objective is to evaluate the safety of PBMT.

The results of this project will support the implementation of PBMT into the standard RD skincare program.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Diagnosis of non-invasive (stage 0) or invasive (stage 1, 2 and 3A) breast adenocarcinoma
* Treatment with primary breast-sparing surgery (lumpectomy) and/or neoadjuvant (preoperative) or adjuvant (postoperative) chemotherapy or hormonal therapy
* Scheduled for postoperative radiotherapy at Ziekenhuis Oost-Limburg, Genk:
* Hypofractionated radiotherapy regimen (i.e. 16 daily fractions of 2.66 Gray to the whole breast followed by a boost of 5 fractions of 2.66 Gray to the tumor bed, 5x/week)

Exclusion Criteria:

* Scheduled for postoperative radiotherapy at Jessa Hospital, Hasselt, Belgium
* Previous irradiation to the same breast
* Metastatic disease
* Concurrent chemotherapy
* Required use of bolus material to deliver radiotherapy (i.e material placed on the to-be- irradiated zone to modulate the delivered dose in order to ensure an optimal distribution of the radiation dose; mostly used for treatment of superficial tumors)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psyschological disorders, dementia, etc. of the participant
* Seizure
* Disorders triggered by lighttake anticoagulants
* Hemorrhagic diatheses
* Pregnancy
* Suspected of carrying serious infectious disease
* HIV positive history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Radiation Dermatitis Grade | week 1
  Objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC) objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | week 2
  Objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC) objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | week 3
  Objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC) objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | week 4
  Objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC) objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | week 5
  Objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC) objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | week 6
  Objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC) objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Assessment | week 1
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Radiation Dermatitis Assessment | week 2
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS 0-4)
Radiation Dermatitis Assessment | week 3
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS 0-4)
Radiation Dermatitis Assessment | week 4
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS 0-4)
Radiation Dermatitis Assessment | week 5
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS 0- 4)
Radiation Dermatitis Assessment | week 6
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS (0 - 4)

SECONDARY OUTCOMES:
Pain evaluation: VAS | week 1
  Patients' pain due to radiodermatitis will be evaluated using the visual analogue scale (VAS 0-10). A VAS is a laminated plastic with descriptors at each end. The patients will be asked to move the sliding marker along the plastic to indicate their subjective experience of pain. Each mark is associated with a certain pain score. A VAS is a well documented, valid, and frequently used measure of pain intensity.
Pain evaluation: VAS | week 2
  Patients' pain due to radiodermatitis will be evaluated using the visual analogue scale (VAS 0-10). A VAS is a laminated plastic with descriptors at each end. The patients will be asked to move the sliding marker along the plastic to indicate their subjective experience of pain. Each mark is associated with a certain pain score. A VAS is a well documented, valid, and frequently used measure of pain intensity.
Pain evaluation: VAS | week 3
  Patients' pain due to radiodermatitis will be evaluated using the visual analogue scale (VAS 0-10). A VAS is a laminated plastic with descriptors at each end. The patients will be asked to move the sliding marker along the plastic to indicate their subjective experience of pain. Each mark is associated with a certain pain score. A VAS is a well documented, valid, and frequently used measure of pain intensity.
Pain evaluation: VAS | week 4
  Patients' pain due to radiodermatitis will be evaluated using the visual analogue scale (VAS 0-10). A VAS is a laminated plastic with descriptors at each end. The patients will be asked to move the sliding marker along the plastic to indicate their subjective experience of pain. Each mark is associated with a certain pain score. A VAS is a well documented, valid, and frequently used measure of pain intensity.
Pain evaluation: VAS | week 5
  Patients' pain due to radiodermatitis will be evaluated using the visual analogue scale (VAS 0-10). A VAS is a laminated plastic with descriptors at each end. The patients will be asked to move the sliding marker along the plastic to indicate their subjective experience of pain. Each mark is associated with a certain pain score. A VAS is a well documented, valid, and frequently used measure of pain intensity.
Pain evaluation: VAS | week 6
  Patients' pain due to radiodermatitis will be evaluated using the visual analogue scale (VAS 0-10). A VAS is a laminated plastic with descriptors at each end. The patients will be asked to move the sliding marker along the plastic to indicate their subjective experience of pain. Each mark is associated with a certain pain score. A VAS is a well documented, valid, and frequently used measure of pain intensity.
Quality of life assessment | week 1
  The Skindex-16 questionnaire will be used to assess patients quality of life. This is the most appropriate questionnaire that accurately and sensitively measures to what extent the patients' life is affected by their skin condition.
Quality of life assessment | week 2
  The Skindex-16 questionnaire will be used to assess patients quality of life. This is the most appropriate questionnaire that accurately and sensitively measures to what extent the patients' life is affected by their skin condition.
Quality of life assessment | week 3
  The Skindex-16 questionnaire will be used to assess patients quality of life. This is the most appropriate questionnaire that accurately and sensitively measures to what extent the patients' life is affected by their skin condition.
Quality of life assessment | week 4
  The Skindex-16 questionnaire will be used to assess patients quality of life. This is the most appropriate questionnaire that accurately and sensitively measures to what extent the patients' life is affected by their skin condition.
Quality of life assessment | week 5
  The Skindex-16 questionnaire will be used to assess patients quality of life. This is the most appropriate questionnaire that accurately and sensitively measures to what extent the patients' life is affected by their skin condition.
Quality of life assessment | week 6
  The Skindex-16 questionnaire will be used to assess patients quality of life. This is the most appropriate questionnaire that accurately and sensitively measures to what extent the patients' life is affected by their skin condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jolien Robijns, PhD, Study Director — Hasselt University
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg Campus St.-Jan, Genk, Limburg
  - Jessa Ziekenhuis, Hasselt